CLINICAL TRIAL: NCT03627390
Title: The Effect of BP-C1 in Treatment of Inoperable Pancreatic Cancer Patients: A Single Centre Pilot Study
Brief Title: BP-C1 in Short-term Treatment of Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meabco A/S (Industry)
Collaborators: Meddoc (Other); Norwegian University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PaCa-BPC1/IIA
Record Dates: First submitted 2018-07-26; First posted 2018-08-13 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Pancreatic Cancer; Unresectable Pancreatic Cancer
Keywords: Benzene polycarboxylic acids complex with cis-diammineplatinum(II); BP-C1; Cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Platinum analogue; Metronomic chemotherapy; Cisplatin; Pancreatic cancer; BP-C2; molybdenum salts of benzene-polycarboxylic acids
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, single center, two arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP-C1 (Experimental): Patients will be treated with BP-C1 for 32 consecutive days
  Interventions: Drug: BP-C1
- BP-C1+BP-C2 (Experimental): Patients will be treated with BP-C1 and BP-C2 for 32 consecutive days
  Interventions: Drug: BP-C1; Drug: BP-C2

INTERVENTIONS:
Drug: BP-C1 — BP-C1, 0.05% solution for injections; doses: 0.035 mg/kg body weight (0.07 mL/kg) intramuscularly once daily for 32 consecutive days
  Other Names: Cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Benzene polycarboxylic acids complex with cis-diammineplatinum(II)
Drug: BP-C2 — BP-C2, 0.15% solution for oral use; 15 ml orally once daily for 32 consecutive days
  Other Names: molybdenum salts of benzene-polycarboxylic acids
  Arms: BP-C1+BP-C2

SUMMARY:
The aim of this study is to investigate the short-term effect and tolerability BP-C1 in patients with metastatic pancreatic cancer who has undergone guideline-recommended chemotherapy.

DETAILED DESCRIPTION:
BP-C1, solution for injections 0.05%, is currently being developed for treatment of patients with metastatic breast cancer and metastatic pancreatic cancer with palliative intent. Active substance of the product, which is a novel platinum-containing anticancer agent developed for intramuscular administration, is a complex between cis-diammineplatinum(II) derived core and an amphiphilic polymer, containing a composition of benzene polycarboxylic acids. The amphiphilic characteristics of the polymer have resulted in a product with clear and significantly altered and improved properties compared to other platinum analogues, e.g. cisplatin, carboplatin and oxaliplatin.

BP-C1 preserves antitumour activity of its predecessors (e.g. cisplatin and carboplatin), additionally offering the following advantages that ensure favourable outcome of treatment in metastatic cancer patients:

* injectable solution (intramuscular) does not cause injection site reactions;
* can be administered at home by a nurse or a patient;
* has an improved pharmacokinetic profile;
* exerts an additional immunomodulatory activity.

BP-C2 is a novel lignin-derived polyphenolic composition with ammonium molybdate. BP-C2, given orally, is believed to reduce the toxicity of chemotherapeutic agents.

This is a single center, two arm, open label pilot study (phase IIa). The eligible patients will be allocated either to BP-C1 arm or to BP-C1+BP-C2 arm and treated for 32 days with further follow-up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders between 18 and 80 years of age with metastatic pancreatic cancer (unresectable pancreatic cancer with increased levels of cancer antigen 19-9), who had an expected survival time of at least 3 months.

Exclusion Criteria:

Patients fulfilling at least one of the following criteria will be excluded from participation in the study:

* Abnormal liver function classified as total bilirubin >136 μmol/L (8.0 mg/dL)
* Abnormal kidney function defined by serum creatinine >120 μmol/L (1.5 mg/dL).
* Abnormal coagulation capacity defined by the relative arbitrary concentration of coagulation factors 2,7,10 < 0.7 or international normalized ratio >1.5.
* Verified metastases to the brain.
* Synchronous cancer except for non-melanoma skin cancer and early stage of cervical cancer.
* Abnormal haematology status defined by hemoglobin < 6.0 g/dL, platelet count < 100,000/mm^3 or leucocytes < 3 x 10^9/L.
* Clinically significant abnormal ECG.
* Karnofsky performance status score <60%.
* Pregnancy or breast-feeding.
* Women of fertile age who do not want to be tested for possible pregnancy.
* Uncontrolled bacterial, viral, fungal or parasite infection.
* Under systemic treatment with corticosteroids or other immunosuppressive drugs in the last 21 days before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals in the last six weeks before start of this trial treatment.
* Not able to understand information.
* Not willing or not able to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2016-03-04 (Actual)

PRIMARY OUTCOMES:
Change (%) in the sum of diameters of target lesions | baseline to Day 32 of treatment
  Diameter of target lesions will be measured by computer tomography (CT) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Maximum Common Toxicity Criteria (CTC) score | baseline to Day 32 of treatment
  Maximum CTC score will be recorded using NCI Common Toxicity Criteria v2.0 divided in 15 categories
Sum CTC score | baseline to Day 32 of treatment
  The Sum CTC score will be a sum of all registered CTC scores by 15 categories

SECONDARY OUTCOMES:
Treatment response | baseline to Day 32 of treatment
  In accordance with RECIST v1.1 the treatment response will be classified as 'complete response', 'partial response', 'stable disease' or 'progressive disease':
  Complete response (CR): disappearance of all target lesions. Partial response (PR): at least 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of diameters.
  Progressive disease (PD): at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum might also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions will also be considered progression.
  Stable disease (SD): neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Scores of the general quality of life cancer questionnaire (EORTC QLQ-C30) | baseline to Day 16 and Day 32 of treatment
  The EORTC QLQ-C30 is a general quality of life questionnaire for cancer patients. The questionnaire contains 30 questions. Three variables will be obtained from the EORTC QLQ-C30: the sum of scores C1 to C5 denoted as "Physical activity problem last week", the sum of scores C6 to C28 denoted as "Discomfort last week", and the sum of scores C29 and C30 denoted as "Health and quality of life"
Number of registered adverse events | screening to Day 32 of treatment and Day 28 of follow-up
  Adverse events (AEs) will be coded according to the MedDRA (version 16.1E). AEs will be systemized by system organ class and by preferred term. AEs will be analyzed by severity, seriousness and relatedness to the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Ibrahim, MD, Principal Investigator — Department of HPH Surgery, National Liver Institute, University of Menoufia, Egypt
Locations (1):
- National Liver Institute, Menoufia University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No